CLINICAL TRIAL: NCT03900962
Title: Effects of Adding Home-based Power Training to a Multidisciplinary Weight Management Service: A Randomised Clinical Trial
Brief Title: Home-based Resistance Training for Adults With Severe Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HullWW2016
Record Dates: First submitted 2019-03-28; First posted 2019-04-03 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Obesity, Morbid
Keywords: Severe obesity; Exercise; Weight management; Resistance training; Power training; Physical function
MeSH Terms: conditions — Obesity, Morbid; Motor Activity

STUDY DESIGN:
Intervention Model Description: After baseline measures were collected, participants were randomly allocated (1:1) to the slow-speed strength training group or the high-speed power training group in block sizes of four using a randomisation sequence created by an independent researcher (GraphPad QuickCalcs, Graphad Software, La Jolla, CA).
Who Masked: Care Provider
Masking Description: The investigator and outcome assessors were not blind to group allocation. It was also not possible to blind participants to the intervention, however, patients were unaware of the study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow-speed strength training (Experimental): The slow-speed strength training group performed the concentric phase of each resistance exercise over two seconds, paused at full extension/flexion for one second, and then performed the eccentric phase for two seconds.
  Interventions: Other: Home-based resistance training; Other: Walking intervention
- High-speed power training (Experimental): During the first three weeks of training, the high-speed power training group completed the concentric phase of each resistance exercise over two seconds, paused at full extension/flexion for one second, and then performed the eccentric phase for two seconds. Thereafter, this group completed the concentric phase of five resistance exercises (squat, press-up, incline chest press, seated row and push-press) as fast as possible whilst still taking two seconds to complete the eccentric phase.
  Interventions: Other: Home-based resistance training; Other: Walking intervention

INTERVENTIONS:
Other: Home-based resistance training — Patients completed two home-based resistance training sessions each week on non-consecutive days for 12 weeks. The programme was delivered online via individual playlists on Youtube (YouTube, San Bruno, California, USA), with each playlist involving an individually-prescribed series of pre-recorded exercise videos. Each session involved a dynamic warm-up followed by 11 resistance exercises using body weight and resistance bands, and finished with static stretching. Participants completed 1-2 sets of 5-12 repetitions at 4-7 on a modified 10-point rating of perceived exertion scale, which corresponded to qualitative descriptors of "moderate" to "hard". Resistance training stimuli were progressed weekly by increasing the external load, modifying the exercise selection, increasing the number of repetitions, and/or increasing the number of sets.
Other: Walking intervention — After the initial baseline assessment, participants recorded the number of steps they walked daily for seven days using a waist-worn pedometer. Participants maintained their usual physical activity levels during this period. Participants were then encouraged to increase their total steps walked each day by 5% each week during the 12-week intervention.

SUMMARY:
This study evaluates whether adding home-based resistance training to a multidisciplinary specialist weight management service can promote weight loss and improve physical function, strength, power and quality of life in adults with severe obesity. The study also investigated whether performing resistance exercises as fast as possible can yield further improvements in physical function compared with traditional slow-speed resistance training.

All recruited participants completed a 3-month home-based resistance training programme with behavioural support; half of the participants performed resistance exercises in a slow and controlled manner, whereas the other half performed resistance exercises with maximal intentional velocity.

DETAILED DESCRIPTION:
Severe obesity reduces muscle contractile function, which manifests as a diminished ability to perform activities of daily living. These functional impairments often lead to pain during movement and a decreased motivation to exercise.

In the United Kingdom (UK), specialist Tier 3 weight management services are provisioned for adults with severe obesity. Tier 3 services comprise a multidisciplinary team (MDT) of specialists and mainly adopt an educational approach, focusing on psychological therapy, dietary modification, pharmacotherapy and physical activity advice. However, current Tier 3 programmes do not specifically address the functional impairments imposed by obesity, which predisposes adults with severe obesity to musculoskeletal pain and pathology.

Adding supervised resistance training to MDT weight management programmes has been shown to improve functional capacity in adults with severe obesity. However, supervised interventions place considerable time and resource burdens on the service provider and patient, which may not be conducive to sustained participation. Obese individuals often report feeling too embarrassed to exercise in front of others and feel uncomfortable appearing in public wearing exercise clothing. Home-based exercise is a convenient alternative to supervised interventions and may promote similar functional adaptations.

Traditional resistance training typically involves sustained contractions at low to moderate velocities. While this method of training is effective for augmenting maximal strength production, which is executed at slow velocities, it may neglect the development of muscle power. This is problematic because lower-limb power has recently emerged as a critical determinant of function in adults with severe obesity.

Power training integrates a high-speed component into conventional resistance training exercises. Research in older adults has consistently shown that power training is superior to conventional slow-speed strength training for improving functionality. Preliminary evidence also exists supporting the superiority of power training in sarcopenic obese adults. Nevertheless, it is unknown whether home-based power training is feasible or effective when added to an MDT weight management programme.

The investigators recruited participants from a UK Tier 3 specialist weight management service. In a prospective, parallel groups, randomised design, participants were randomly allocated to a slow-speed strength training group or a high-speed power training group. Both groups completed a 12-week, individualised, home-based resistance training intervention (2x/week) with behavioural support. The high-speed power training group performed resistance exercises with maximal intended concentric velocity whereas the slow-speed strength training group maintained a slow (2-s) lifting speed. Outcomes were assessed at baseline, 3-month (post-intervention), and 6-month (follow-up) endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a Tier 3 specialist weight management service in the United Kingdom
* Body mass index of ≥ 40 kg/m2 or between 35 and 40 kg/m2 with a serious co-morbidity (such as type 2 diabetes or obstructive sleep apnoea).
* Aged ≥ 18 years
* Willing and able to give written informed consent.
* Understand written and verbal instructions in English

Exclusion Criteria:

* Unstable chronic disease state
* Prior myocardial infarction or heart failure
* Poorly controlled hypertension (≥ 180/110 mmHg)
* Uncontrolled supraventricular tachycardia (≥ 100 bpm)
* Absolute contraindications to exercise testing and training as defined by the American College of Sports Medicine
* Current participation in a structured exercise regime (≥ 2x/week for the last 3 months)
* Body mass ≥ 200 kg
* Any pre-existing musculoskeletal or neurological condition that could affect their ability to complete the training and testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Lower-limb power (W) | 3-month endpoint
  Mean power was measured in the sit-to-stand transfer with a wearable inertial sensor (PUSH, PUSH Inc., Toronto, Canada). The device is worn on the participant's forearm and measures acceleration in the upwards phase of the movement. Power is then calculated as velocity x force, where velocity is the integral of acceleration, and force is the product of mass and acceleration. The test was administered in a firm bariatric chair (height, 48 cm; depth, 56 cm; width, 69 cm). From a seated position, participants were instructed to maintain their arms crossed against their chest and stand up as quickly as possible (legs straight), before returning back to the initial seated position in a controlled manner (full weight on chair). Two warm-up trials were performed, followed by three repetitions separated by 60 seconds of rest. Additional trials were performed if the arms moved away from the chest.

SECONDARY OUTCOMES:
Number of recruited participants | During the 13-month recruitment period
  Measured as the number of eligible participants who were eligible and consented to participate in the trial. This will be reported in a Consolidated Standards of Reporting Trials (CONSORT) participant flowchart.
Number of adverse events | During the 3-month intervention period
  The number of adverse events were recorded to determine the feasibility of the exercise intervention. An adverse event was defined as the occurrence of any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the exercise intervention. The type of adverse events was also noted.
Attrition rate | During the 3-month intervention period
  Established as the number of patients who discontinued the exercise intervention.
Number of patients lost to follow-up | 3-month and 6-month endpoints
  Participants lost to follow-up were characterised as those who completed the exercise intervention but did not complete endpoint testing.
Number of exercise sessions completed | During the 3-month intervention period
  The number of exercise sessions completed by each participant was recorded. The maximum number of exercise sessions that participants could complete was 24, so adherence ranged from 0 to 24 sessions, with higher scores indicating greater adherence.
Body mass (kg) | 3-month and 6-month endpoints
  A calibrated digital scale (seca 813, SECA, Birmingham, UK) was used to measure body mass to the nearest 0.1 kg. Participants wore light clothing and removed their footwear before stepping on the scale.
Waist and hip circumference (cm) | 3-month and 6-month endpoints
  Using a non-stretching measuring tape (seca 201, SECA, Birmingham, UK), waist and hip circumferences were measured to the nearest 0.1 cm. Participants stood upright with their hands by their side and feet positioned shoulder-width apart. The waist circumference measurement was made at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest at the end of a normal expiration. Hip circumference was taken around the widest portion of the buttocks.
Waist to hip ratio | 3-month and 6-month endpoints
  Waist circumference (cm) was divided by hip circumference (cm) to calculate the waist to hip ratio.
Six-minute walk test (m) | 3-month and 6-month endpoints
  Participants were instructed to walk at their own maximal pace back and forth along a flat 30 m surface, covering as much ground as they could in six minutes. All instructions, encouragement and monitoring adhered to the guidelines provided by the American Thoracic Society (ATS, 2002).
Timed up-and-go (s) | 3-month and 6-month endpoints
  Participants sat in a firm bariatric chair and were instructed to stand up, walk three metres before turning 180° around a cone and returning to the chair to sit down.
30-s chair sit-to-stand test (s) | 3-month and 6-month endpoints
  The test was administered in a firm bariatric chair, which was supported against a wall. Participants began seated and were subsequently instructed to rise to a full standing position (legs straight) and then return to the seat (full weight on chair) with both arms crossed against the chest. A practice trial of two repetitions was given to check correct form, followed by one test trial.
Shoulder press and seated row one repetition maximums (kg) | 3-month and 6-month endpoints
  Shoulder press and seated row one repetition maximum (1RMs) were determined with resistance machines (Life Fitness, Ely, Cambridgeshire, UK). Participants performed five repetitions at 3 rating of perceived exertion (RPE) ("easy"), three repetitions at 5 RPE ("somewhat hard"), and two repetitions at 8 RPE ("very hard"). Thereafter, the load was progressively increased (2.5-5kg) until the participant could not complete a repetition using correct technique through a full range of motion. The last successful attempt was taken as the 1RM.
Lower-limb power (W) | 6-month endpoint
  Mean power was measured in the sit-to-stand transfer with a wearable inertial sensor. The device is worn on the participant's forearm and measures acceleration in the upwards phase of the movement. Power is then calculated as velocity x force, where velocity is the integral of acceleration, and force is the product of mass and acceleration. The test was administered in a firm bariatric chair. From a seated position, participants were instructed to maintain their arms crossed against their chest and stand up as quickly as possible (legs straight), before returning back to the initial seated position in a controlled manner (full weight on chair). Two warm-up trials were performed, followed by three repetitions separated by 60 seconds of rest. Additional trials were performed if the arms moved away from the chest.
Lower-limb movement velocity (m/s) | 3-month and 6-month endpoints
  Mean velocity was calculated in the sit-to-stand movement using a wearable inertial sensor.
Shoulder press velocity (m/s) | 3-month and 6-month endpoints
  Participants lifted 50% of the load achieved in the 1RM test as fast as possible. Two warm-up trials were performed, followed by three repetitions separated by 60 seconds of rest. A wearable inertial sensor was used to measure mean velocity in the concentric phase of each repetition.
Shoulder press power (W) | 3-month and 6-month endpoints
  Participants lifted 50% of the load achieved in the 1RM test as fast as possible. Two warm-up trials were performed, followed by three repetitions separated by 60 seconds of rest. A wearable inertial sensor was used to measure mean power in the concentric phase of each repetition.
EuroQol 5-level questionnaire (EQ-5D-5L) | 3-month and 6-month endpoints
  The EQ-5D-5L is a generic, self-administered measure of health-related quality of life that gathers descriptive information on five main dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The participant indicates the level that best describes their state of health on that day. This results in a 1-digit number expressing the level selected for that dimension, which were combined to produce a five-digit number describing the participant's health status (ranging from 11111 to 55555). This is then converted to a single index value based on the EQ-5D-5L Crosswalk value set for England that ranges from -0.594 (worst possible health) to 1.000 (best possible health).
EuroQoL visual analogue scale (EQ-VAS) | 3-month and 6-month endpoints
  The EQ-VAS is a single-item measure of overall health that has demonstrated acceptable psychometric properties in several populations. The participant rates their current perceived health status on a 20 cm, vertical visual analogue scale that ranges from 0 ("The worst health you can imagine") to 100 ("The best health you can imagine"). Higher scores indicate a better health status.
Obesity and Weight Loss Quality of Life Instrument (OWLQOL) | 3-month and 6-month endpoints
  The OWLQOL measured obesity-specific quality of life, which is self-administered and contains 17-items that explore unobservable needs such as freedom from stigma and attainment of culturally appropriate goals. Each item has a 7-point Likert-like response scale ranging from 0 ("Not at all") to 6 ("A very great deal"). The raw score is transformed to a standardised scale of 0 to 100, where higher scores indicate better quality of life.
Weight-related symptom measure (WRSM) | 3-month and 6-month endpoints
  The WRSM is a 20-item, self-report measure for the presence and bothersomeness of obesity symptoms. Participants responded either "yes" or "no" as to whether they experienced the symptom in the last four weeks and then rated the degree of bothersomeness that having the symptom caused them. The bothersomeness options are on a 7-point Likert-like response scale ranging from 0 ("Not at all") to 6 ("A very great deal"). A total score is calculated by adding up all the bothersomeness scores for each symptom. Scores range from 0 to 120, with higher scores indicating a higher or worse experience of symptoms.
Sessional heart rate (%) | During the 3-month intervention period
  Participants recorded their average heart rate, maximum heart rate using their heart rate monitor (FT1, Polar Electro, Kempele, Finland). Recording commenced before the start of the warm-up and stopped immediately after the last resistance exercise (before the cool-down). Heart rate was expressed as a percentage of heart rate reserve.
Session duration (minutes) | During the 3-month intervention period
  Participants recorded the duration of each session using their heart rate monitor. Recording commenced before the start of the warm-up and stopped immediately after the last resistance exercise (before the cool-down).
Total number of repetitions during each resistance training session | During the 3-month intervention period
  The total number of repetitions performed during each resistance training session was calculated as: number of sets x number of exercises x number of repetitions in each exercise.
Step count | During the 3-month intervention period
  Participants recorded the number of steps they walked daily using a waist-worn pedometer. Steps counts are reported as the average number of daily steps performed during each week
Isometric mid-thigh pull (kg) | 3-month and 6-month endpoints
  Using an analogue back dynamometer (Takei Scientific Instruments Co. Ltd., TKK 5002 Back-A, Tokyo, Japan), participants maximally extended their knees and trunk for five seconds without bending their back. The height of the handle was individually adjusted so that the bar rested midway up the thigh and there was 145° of knee flexion, which was measured with a handheld goniometer (Economy Jamar Goniometer, JAMAR Technologies, Inc., Hatfield, Pennsylvania, USA). Two trials were performed with a two-minute rest period in between. Each trial was recorded to the nearest 1 kg, with the maximum value used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca V Vince, PhD, Principal Investigator — University of Hull

IPD SHARING:
Plan to Share IPD: Yes
All raw data and imputed data will be made available via the open science framework (https://osf.io/)
Supporting Information: SAP, Analytic Code
Time Frame: Immediately after publication
Access Criteria: Raw data will be made available to the public without restriction.

REFERENCES:
- [Background] Ling C, Kelechi T, Mueller M, Brotherton S, Smith S. Gait and Function in Class III Obesity. J Obes. 2012;2012:257468. doi: 10.1155/2012/257468. Epub 2012 Feb 16. PMID 22496967
- [Background] Shultz SP, Byrne NM, Hills AP. Musculoskeletal Function and Obesity: Implications for Physical Activity. Curr Obes Rep. 2014 Sep;3(3):355-60. doi: 10.1007/s13679-014-0107-x. PMID 26626767
- [Background] Brown TJ, O'Malley C, Blackshaw J, Coulton V, Tedstone A, Summerbell C, Ells LJ. Exploring the evidence base for Tier 3 weight management interventions for adults: a systematic review. Clin Obes. 2017 Oct;7(5):260-272. doi: 10.1111/cob.12204. Epub 2017 Jul 10. PMID 28695579
- [Background] Herring LY, Wagstaff C, Scott A. The efficacy of 12 weeks supervised exercise in obesity management. Clin Obes. 2014 Aug;4(4):220-7. doi: 10.1111/cob.12063. Epub 2014 Jun 26. PMID 25826793
- [Background] Baillot A, Mampuya WM, Comeau E, Meziat-Burdin A, Langlois MF. Feasibility and impacts of supervised exercise training in subjects with obesity awaiting bariatric surgery: a pilot study. Obes Surg. 2013 Jul;23(7):882-91. doi: 10.1007/s11695-013-0875-5. PMID 23430477
- [Background] Wiklund M, Olsen MF, Willen C. Physical activity as viewed by adults with severe obesity, awaiting gastric bypass surgery. Physiother Res Int. 2011 Sep;16(3):179-86. doi: 10.1002/pri.497. Epub 2010 Nov 9. PMID 21061456
- [Background] Orange ST, Marshall P, Madden LA, Vince RV. Short-Term Training and Detraining Effects of Supervised vs. Unsupervised Resistance Exercise in Aging Adults. J Strength Cond Res. 2019 Oct;33(10):2733-2742. doi: 10.1519/JSC.0000000000002536. PMID 29528961
- [Background] Orange ST, Marshall P, Madden LA, Vince RV. Can sit-to-stand muscle power explain the ability to perform functional tasks in adults with severe obesity? J Sports Sci. 2019 Jun;37(11):1227-1234. doi: 10.1080/02640414.2018.1553500. Epub 2018 Dec 5. PMID 30517830
- [Background] Steib S, Schoene D, Pfeifer K. Dose-response relationship of resistance training in older adults: a meta-analysis. Med Sci Sports Exerc. 2010 May;42(5):902-14. doi: 10.1249/MSS.0b013e3181c34465. PMID 19996996
- [Background] Tschopp M, Sattelmayer MK, Hilfiker R. Is power training or conventional resistance training better for function in elderly persons? A meta-analysis. Age Ageing. 2011 Sep;40(5):549-56. doi: 10.1093/ageing/afr005. Epub 2011 Mar 7. PMID 21383023
- [Background] Balachandran A, Krawczyk SN, Potiaumpai M, Signorile JF. High-speed circuit training vs hypertrophy training to improve physical function in sarcopenic obese adults: a randomized controlled trial. Exp Gerontol. 2014 Dec;60:64-71. doi: 10.1016/j.exger.2014.09.016. Epub 2014 Oct 1. PMID 25281504
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Orange ST, Metcalfe JW, Liefeith A, Marshall P, Madden LA, Fewster CR, Vince RV. Validity and Reliability of a Wearable Inertial Sensor to Measure Velocity and Power in the Back Squat and Bench Press. J Strength Cond Res. 2019 Sep;33(9):2398-2408. doi: 10.1519/JSC.0000000000002574. PMID 29742745

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT03900962/SAP_000.pdf